CLINICAL TRIAL: NCT00747643
Title: Varenicline Effects on Cue Reactivity and Smoking Reward/Reinforcement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: MCC-15444; 106842 (Other: USF IRB)
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Results first posted 2011-11-29 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2011-10

CONDITIONS: Tobacco Dependence
Keywords: tobacco; nicotine; smoking; reward; reinforcement; craving; cues; conditioned stimuli; cue reactivity
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Active Comparator): For participants in the varenicline group, the medication doses followed the recommended dose schedule for the first 15 days of treatment: 0.5 mg once a day on days 1-3, 0.5 mg twice a day on days 4-7, and 1 mg twice a day on days 8-15.
  Interventions: Drug: varenicline
- Placebo (Placebo Comparator): Participants in this group received a placebo instead of medication. The placebo was taken once a day on days 1-3, twice a day on days 4-15.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — Participants in this group received varenicline according to the schedule in the Arm Description.
  Other Names: Chantix™
  Arms: Varenicline
Drug: placebo — Participants in this group received a placebo and did not receive any active medication according to the schedule in the Arm Description.
  Arms: Placebo

SUMMARY:
The purpose of this study was to find out how varenicline works to help people quit smoking. Varenicline, also known as Chantix™, is an U.S. Food and Drug Administration (FDA) approved medication that has been shown to help people quit smoking. This study was trying to evaluate whether varenicline would change the response to smoking and the desire for cigarettes when compared to an inactive placebo control. This was not a quit smoking treatment study, and participants were not asked or required to stop smoking while in this study.

DETAILED DESCRIPTION:
We proposed the following primary hypotheses:

1. Tonic (i.e., non-cue-provoked) craving levels would be lower in participants receiving varenicline versus placebo.
2. Cue-provoked cravings (self-report and physiological responding) would be lower in participants receiving varenicline versus placebo. (Secondary indices of craving include heart rate and skin conductance.)
3. The two primary indices of nicotine reward/reinforcement (mCEQ and choice index) would be lower in participants receiving varenicline versus placebo. (Secondary indices of nicotine reinforcement include smoking topography variables.)

A final sample of 100 non-treatment seeking daily smokers were recruited from the Tampa-St. Petersburg-Clearwater Metropolitan Area via paid advertisements in, and press releases to, local newspapers, as well as targeted outdoor advertising via flyers (e.g., on public transportation).

Following the screening session, participants were randomly assigned to receive either varenicline or placebo medication.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* Smoke at least 15 cigarettes daily
* Expired-air carbon monoxide (CO) > 10 ppm
* Medically eligible to receive Varenicline.

Exclusion Criteria:

* Patients who are pregnant or lactating
* Who show evidence of renal dysfunction (BUN > 25 mg/dL, or creatinine > 1.3 mg/dL)
* Are using other smoking cessation medications
* Have current psychiatric disorders (i.e. major depression, manic depression, and/or psychotic episodes) as determined by the Structured Clinical Interview for DSM Disorders (SCID) (First et al., 1996), will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2008-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brandon, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To achieve a sample size of 100 following attrition, we screened 573 smokers from the community and randomized 100 non-treatment seeking daily smokers to the two conditions. Smokers who were using other smoking cessation medications, or who had current mood or psychotic disorders were excluded.
Pre-assignment Details: Participants completed a baseline evaluation including screening for inclusion and exclusion criteria, a medical evaluation, basic metabolic panel and pregnancy test for females. Participants who met all of the inclusion criteria were scheduled for the assessment sessions.
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 82 | 81
Completed | 46 | 54
Not Completed | 36 | 27
Not completed — Withdrawal by Subject | 36 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 46 | 54 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 54 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 28 | 33 | 61
Region of Enrollment [Number; unit: participants]
  United States | 46 | 54 | 100

OUTCOME MEASURES:

1. Primary Outcome: Tonic Craving Score (QSU) Based on Self Reports
Description: Tonic Craving 1 (lowest) to 7 (highest). The Questionnaire of Smoking Urges (QSU), our primary measure of tonic craving, is a 32-item instrument, including 2 separate factor scales that roughly correspond to the desire to smoke for its pleasurable effects (positive reinforcement) or to remove unpleasant feelings of negative affect or withdrawal (negative reinforcement) (Tiffany and Drobes 1991). Following overnight abstinence, each session included assessment of tonic craving, reactivity (including craving) to smoking cues.
Time Frame: 3 weeks per participant
Population: Per Protocol
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 46 | 54
Scores on a scale | 3.53 (.21) | 4.93 (.19)

2. Secondary Outcome: Smoking Topography - Number of Puffs on a Cigarette
Description: # Puffs = total number of puffs taken at Assessment Session.
Time Frame: 3 weeks per participant
Population: Per Protocol
Measure: Mean (Standard Error); unit: Puffs on a Cigarette
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 46 | 54
Puffs on a Cigarette | 6.05 (.77) | 9.86 (.76)

3. Primary Outcome: Cue-provoked Cravings
Description: Strength of Craving 0 (lowest) to 20 (highest). One item 0 - 20 Likert scale "How strong was your craving to smoke a cigarette?"
Time Frame: 3 weeks per participant
Population: Per Protocol
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 46 | 54
Scores on a scale | 11.18 (.76) | 14.61 (.69)

4. Secondary Outcome: A Measure of the Subjective Expected Value of a Cigarette
Description: The cigarette choice procedure (Kidorf, Stitzer, and Griffiths, 1995) is a measure of the desire to smoke a cigarette. Participants are asked to hypothetically choose between smoking a cigarette now or receiving a small amount of money (from 10 cents up to $6 in increments of 10 cents). A crossover ($) value, at and above which participants prefer money, is obtained (Reid, Palmar, Raghavan, and Flammino, 2007).
Time Frame: 3 weeks per participant
Population: Per Protocol
Measure: Mean (Standard Error); unit: Dollars
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 46 | 54
Dollars | 2.46 (.30) | 3.72 (.28)

ADVERSE EVENTS:
Time Frame: 3 weeks per participant
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/81
Other Adverse Events (participants affected / at risk) | 0/82 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No